CLINICAL TRIAL: NCT06935448
Title: Effect of an Enhanced Recovery After Surgery Program on Outcomes After Pancreatoduodenectomy; Experience From Two Referral Centers in Central Greece.
Brief Title: Effect of an Enhanced Recovery After Surgery Program on Outcomes After Pancreatoduodenectomy
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DESPOINA LIOTIRI, Dr, University of Thessaly
Other Study IDs: UNIVERSITY OF THESSALY 2412
Record Dates: First submitted 2025-04-08; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pancreatectomy; Enhanced Recovery After Surgery; Pancreatic Cancer Resectable
Keywords: pancreatectomy; enhanced recovery after surgery; pancreatic cancer resectable; outcomes research
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: traditional perioperative care
- ERAS group: enhanced recovery after surgery perioperative care
  Interventions: Other: enhanced recovery after surgery

INTERVENTIONS:
Other: enhanced recovery after surgery — ERAS group follows the enhanced recovery after surgery program which involves 20 elements
  Groups: ERAS group

SUMMARY:
This study assesses whether patients with pancreatic cancer who undergo surgery experience improved outcomes following the implementation of a multidisciplinary care pathway, specifically an enhanced recovery after surgery (ERAS) program.

This pathway includes various interventions in the preoperative, intraoperative, and postoperative care of these patients, all aimed at enhancing their health status and postoperative results.

DETAILED DESCRIPTION:
This prospective observational study is conducted by the same surgical team at two high-volume pancreatic cancer referral centers in Greece.

Patients undergoing elective pancreatic surgery are prospectively enrolled and managed according to a standardized ERAS protocol (ERAS group).

A control group, which received standard perioperative care before the implementation of ERAS, was retrospectively selected and matched based on demographic and clinical parameters.

The primary study endpoint is the length of hospital stay (LOS), while secondary endpoints include 30-day mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnosis of pancreatic cancer
* elective open pancreatic surgery

Exclusion Criteria:

* age <18 years
* emergency pancreatic surgery
* other surgical procedures
* missing data
* lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreatic surgery in two pancreatic cancer referral centers in central Greece, namely the University Hospital of Larissa, and IASO Thessalias general hospital
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
impact on length of stay | within 30 days of surgery
  total number of days spent in the hospital including any readmission

SECONDARY OUTCOMES:
impact on overall morbidity | within 30 days from surgery
  number of any perioperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: DESPOINA LIOTIRI, MD, DESAIC, EDRA, MSc, PhD(c), Principal Investigator — University of Thessaly; ATHINA SAMARA, MD, MSc, PhD(c), Principal Investigator — University of Thessaly; NIKOLAOS BEIS, MD, Principal Investigator — University of Thessaly; DIMITRIS ZACHAROULIS, PROFESSOR OF SURGERY, Study Chair — University of Thessaly; Alexandros Diamantis, MD, MSc, PhD, Principal Investigator — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Cardini B, Primavesi F, Maglione M, et al. Outcomes following pancreatic resections-results and challenges of an Austrian university hospital compared to nationwide data and international centres. Eur Surg (2019) 51:81-89. https://doi.org/10.1007/s10353-019-0585-x
- [Background] Lau CS, Chamberlain RS. Enhanced Recovery After Surgery Programs Improve Patient Outcomes and Recovery: A Meta-analysis. World J Surg. 2017 Apr;41(4):899-913. doi: 10.1007/s00268-016-3807-4. PMID 27822725
- See also: ERAS society guidelines for pancreatic surgery — https://erassociety.org/guidelines/